CLINICAL TRIAL: NCT07127809
Title: A Multilevel Study on the Effects of a Mindfulness-Based Intervention Targeting Psychological Capital on Job Burnout Among Nurses: A Randomized Controlled Trial
Brief Title: Mindfulness-Based Intervention Targeting Psychological Capital to Reduce Job Burnout Among Nurses
Acronym: MINCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taizhou Hospital (Other)
Collaborators: Taizhou University (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Mengjie Xia, Lecturer in Nursing, Taizhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25EZC07
Record Dates: First submitted 2025-07-18; First posted 2025-08-17 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Burnout; Psychological Capital; Mental Health; Mindfulness-based Intervention
Keywords: Job burnout; Mindfulness-based intervention; Psychological capital; Multilevel analysis
MeSH Terms: conditions — Burnout, Psychological; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Practice (Experimental): Nurses receive structured mindfulness practice in addition to routine work.
  Interventions: Behavioral: Mindfulness Practice
- Control Group (No Intervention): Nurses continue routine work without additional intervention.

INTERVENTIONS:
Behavioral: Mindfulness Practice — Participants in this group will engage in a structured mindfulness practice program delivered via a custom-developed mobile app. The intervention includes guided mindfulness exercises such as meditation, breathing techniques, and body awareness, designed to be practiced daily alongside routine nursing duties. The program aims to enhance psychological capital and reduce job burnout symptoms over a 40-day intervention period, with follow-up assessments at 2 and 4 months post-intervention.
  Arms: Mindfulness Practice

SUMMARY:
The goal of this clinical trial is to evaluate whether a mindfulness-based intervention can reduce job burnout and enhance psychological capital among hospital nurses. The study will involve female nurses aged 22-50 working in four tertiary hospitals in Taizhou, China.

The main questions it aims to answer are:

Can mindfulness practice improve nurses' psychological capital (as measured by the Psychological Capital Questionnaire, PCQ-24)? Can it reduce job burnout (as measured by the Maslach Burnout Inventory - General Survey, MBI-GS)? Is there a sustained effect over time (2 and 4 months post-intervention)?

Researchers will compare the intervention group (mindfulness practice) with a control group (routine work, no additional intervention) to see if mindfulness leads to measurable improvements in psychological well-being and burnout symptoms.

Participants will:

Complete online questionnaires at baseline,and at 2 and 4 month follow-ups. Engage in a structured mindfulness practice program delivered via a mobile app (intervention group only).

Continue their routine work responsibilities throughout the study period.

This study also explores the influence of multilevel psychological capital-at the individual, organizational, and family levels-on nurse burnout, aiming to develop an evidence-based, scalable approach to address nurse mental health in high-stress healthcare environments.

DETAILED DESCRIPTION:
This randomized controlled trial aims to assess the effectiveness of a mindfulness-based intervention in reducing job burnout among nurses by enhancing their psychological capital. The study adopts a multilevel perspective, examining how individual, organizational (nurse managers), and family (relatives) psychological capital influence nurse burnout.

A total of 1030 participants-including nurses, head nurses, and family members-will complete baseline assessments. Among them, 124 nurses with moderate to high burnout levels will be randomly assigned to either a mindfulness intervention group or a control group. The intervention will be delivered via a mobile app and integrated into nurses' daily routines.

Outcomes will be measured at multiple time points using validated tools: Psychological Capital Questionnaire (PCQ-24), Maslach Burnout Inventory - General Survey (MBI-GS), and Five Facet Mindfulness Questionnaire (FFMQ). This study will explore both immediate and long-term intervention effects and aims to develop a scalable model for burnout prevention among healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurses aged 22-50
* Employed full-time in tertiary hospitals in Taizhou, China
* Moderate or high levels of burnout (Maslach Burnout Inventory - General Survey screening)
* Provided informed consent

Exclusion Criteria:

* Diagnosed psychiatric disorders or ongoing psychotropic medication
* Prior formal mindfulness training
* Inability to use mobile applications

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Job Burnout Level measured by the Maslach Burnout Inventory - General Survey (MBI-GS) | Baseline, Day 40, and 2- and 4-month follow-ups
  Evaluate the change in job burnout symptoms (emotional exhaustion, cynicism, and reduced professional efficacy) among nurses in the intervention group compared to control.
Psychological Capital Level measured by the Psychological Capital Questionnaire (PCQ-24) | Baseline, Day 40, and 2- and 4-month follow-ups
  Assess the change in psychological capital, including self-efficacy, hope, resilience, and optimism among nurses receiving the mindfulness intervention compared to control.

SECONDARY OUTCOMES:
Mindfulness Level measured by the Five Facet Mindfulness Questionnaire (FFMQ) | Baseline, Day 40, and 2- and 4-month follow-ups
  Measure changes in mindfulness traits (observing, describing, acting with awareness, non-judging, non-reactivity) following the mindfulness intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Taizhou central hospital, Taizhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including the final dataset and accompanying data dictionary, will be made available to researchers outside the primary study group.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be available beginning 12 months after publication of the primary results and for a period of 5 years thereafter.
Access Criteria: Qualified researchers may request access by contacting the principal investigator at xiamengjie@tzc.edu.cn. Requests must include a methodologically sound research proposal and will require signing a data use agreement. Data will be shared via a secure, password-protected repository.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-18): https://cdn.clinicaltrials.gov/large-docs/09/NCT07127809/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT07127809/ICF_001.pdf